CLINICAL TRIAL: NCT06296524
Title: Effect of Footcore Exercises on Navicular Drop and Plantar Pressure Distribution in Asymptomatic Individual With Flatfoot: A Pilot RCT
Brief Title: Effect of Footcore Exercises on Navicular Drop and Plantar Pressure Distribution in Asymptomatic Individual With Flatfoot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Subhasish Chatterjee, Clinical Professor, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPC-2022-09
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Flatfoot
Keywords: Footcore, Harris Mat, Plantar pressure.
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Footcore exercises and conventional therapy (Experimental): Participants received Footcore exercises along with conventional therapy for 4 weeks, twice a day Footcore exercises includes toe yoga, toe spreads, foot doming, calf stretch, ball rolling. + conventional therapy
  Interventions: Other: Footcore exercises and conventional therapy
- Conventional Therapy (Active Comparator): Participants received conventional physiotherapy treatment, which includes toe curl, picking of small object, heel raise (For 4 weeks, twice a day).
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Footcore exercises and conventional therapy — 30 minutes exercises protocol will be provided
  Arms: Footcore exercises and conventional therapy
Other: conventional therapy — conventional therapy will be provided.
  Arms: Conventional Therapy

SUMMARY:
Pes Planus is a medical condition in which arch of the foot is flattened, causing the entire sole of the foot to contact the floor. For those with flat feet, footcore exercises might be an effective non-invasive therapy. Footcore exercises aim to strengthen the intrinsic foot muscles that maintain the foot arch, enhance foot function and reduce the risk of injury in persons with flatfoot.

DETAILED DESCRIPTION:
A pilot, random research with 10 participants was undertaken. Two groups, Experimental group and Control group, were randomly selected among the subjects. Participant completed the informed consent form before the navicular drop test and Harris Mat was used to measure the foot pressure. Footcore exercises and conventional therapy was given for four weeks ,twice a day for 6 days. While the Control group just received conventional treatment, the Experimental group combined Footcore exercise with it. The data will be analyzed using SPSS 26.0 software.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals having flat feet.
2. those with a height difference of ≥ 10 mm during the navicular drop test.
3. No history of foot or ankle surgery.

Exclusion Criteria:

1. Any lower limb injury
2. Healing fracture of lower limb33
3. Any neuromuscular disorder 25
4. Recent surgery
5. Any open wound.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Navicular Drop Test | 1 month
  A thick, white index card was used for the navicular drop test, which measured the navicular height. The card was positioned from the surface in a vertical position, passing the navicular bone, on the medial portion of the hindfoot, parallel to the subject's feet (kept in a subtalar neutral position). The floor was measured while sitting and standing, and the level of the navicular tubercle's highest point was marked on the card.An increased intra- (ICC = 0.73-0.96) and inter-rater reliability (ICC = 0.92) along with significant Pearson correlations to radiographic images (r = 0.89-0.92)
  have been shown when the NDT was modified to address these issues using the Sit-to-Stand Navicular Drop Test (SSNDT) method with digital photographs.
Harris Mat for Plantar Pressure Distribution | 1 month
  On a Harris-Beth mat, the patients' footprints were captured . Each foot's static imprint was captured while the body was supported by just half of its weight. The broadest region of the arch and the heel of each foot were measured, and the arch index and foot pressure for both feet were determined by dividing the former value by the latter, as explained by Staheli et al.Interrater and interrater reliability of the footprint parameters both revealed ICC values close to or greater than 0.9. Previous research found that the SI and CSI have great reliability (0.914-0.998)

CONTACTS AND LOCATIONS:
Overall Officials: Mousumi Saha, MPT, Principal Investigator — MMIPR
Locations (1):
- MMIPR, Ambāla, Haryana, India